CLINICAL TRIAL: NCT02890498
Title: Vaginal Microbiota as a Decisive Factor in Vaginal Prosthetic Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2016/RdT-02
Record Dates: First submitted 2016-08-26; First posted 2016-09-07 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-08

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
Retrospective analysis of vaginal microbiota in the post-operative course of patient operated for genital prolapse with vaginal mesh with or without mesh related complication

DETAILED DESCRIPTION:
We propose to collect vaginal specimens to obtain exfoliated mucosal cells from women who had vaginal mesh implantation for POP complicated by mesh erosion into the vagina (cases).

We aim to recruit women who will receive exactly the same clinical investigations (outlined below), follow up and management.

Samples from patients without complications after mesh surgery will be used as controls since there are ethical difficulties in obtaining cold-cup swabs from 'normal' women and cystoscopy for conditions other than OAB or USI in premenopausal women is rare.

Both cases and controls will be identified by the urogynaecology team based on surgical outcome reports and follow-up documentation. Cases and controls will be invited to participate by the research team. Relevant members of the research team (Dr Nikolaus Veit-Rubin, Pr Renaud DeTayrac, and Mr Vikram Khullar) have extensive experience in urogynaecological investigation and pelvic floor assessment.

Cases and controls will be provided with an information leaflet about the study and will be asked to sign informed consent for the biopsies and a high vaginal swab will be taken. Consent will be taken either a trained member of the urogynaecology team. All participants will complete the 'P-QoL Questionnaire" for symptoms relative to POP. Clinical assessment will include a comprehensive relevant past medical history, calculation of BMI, urinalysis, standardized POP-Q Quantification and abdominal examination.

Specimens collected to be analysed will be a high vaginal swab following fully informed written consent. The specimens of Vaginal swab will be processed to extract and purify the DNA and then the exact bacterial genomic make up will be sequenced and analysed to identify the exact species of bacteria within the samples. Further detailed protocol of the mentioned procedures is outlined in the attached protocol.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 and over who have consented for vaginal mesh surgery for pelvic organ prolapse at the the Nîmes University Hospital, France

Exclusion Criteria:

* Pregnant or breast feeding
* Unwilling or unable to complete questionnaire or give valid consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females aged 18 and over who have consented for vaginal mesh surgery for pelvic organ prolapse at the Nîmes University Hospital, France
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Microbiota diversity (Shannon's H index) | Day 0